CLINICAL TRIAL: NCT07312188
Title: A Phase II Study of F182112 Combined With Different Administration Regimens in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of F182112 in the Treatment of Patients With Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NTP-F182112-101
Record Dates: First submitted 2025-04-24; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- F182112 combined with different administration regimens (Experimental): F182112 combined with different administration regimens
  Interventions: Drug: F182112+P; Drug: F182112+CD38

INTERVENTIONS:
Drug: F182112+P — F182112 + P
  Other Names: F182112; Pomalidomide
Drug: F182112+CD38 — F182112+CD38
  Other Names: F182112; BCMA CD3; CD38 monoclonal antibody

SUMMARY:
This is a single - arm, multi - cohort, open - label, multi - center Phase II clinical study. It aims to evaluate the efficacy and safety of F182112 combined with different administration regimens in patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
The study plans to enroll approximately 90 patients with relapsed or refractory multiple myeloma at around 20 study centers.

Primary objective:

The objective response rate (ORR) of F182112 combined with different administration regimens in patients with relapsed or refractory multiple myeloma.

Secondary objective:

The efficacy of F182112 combined with different administration regimens in patients with relapsed or refractory multiple myeloma (complete response rate [CRR], progression - free survival [PFS], overall survival [OS], duration of response [DOR], time to response [TTR], time to progression [TTP], minimal residual disease - negative rate); The incidence and grade of adverse events (AE), serious adverse events (SAE), abnormal laboratory test indicators.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with multiple myeloma according to the IMWG 2016 criteria.
* The previous treatment regimen must contain lenalidomide (lenalidomide must be used continuously for at least 2 cycles) and a proteasome inhibitor.
* Participants whose previous treatment regimen contained pomalidomide or who were intolerant to pomalidomide cannot be enrolled.
* Have an ECOG performance status score of 0 - 2.
* Meet at least one of the following measurable disease indicators:

  1. Serum M - protein ≥ 5 g/L.
  2. Urine M - protein ≥ 200 mg/24 h.
  3. Serum free light chain (FLC) test: Involved FLC level ≥ 100 mg/L and abnormal serum free light chain ratio (< 0.26 or > 1.65).

Exclusion Criteria:

* Patients with primary light - chain amyloidosis or plasma cell leukemia .
* Patients with symptoms of central nervous system involvement of multiple myeloma.
* Patients with a history of other malignancies other than multiple myeloma within 3 years before the first dose.
* Patients with active mucosal or visceral bleeding.
* Patients who have previously received BCMA - targeted therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2028-05-20 (Estimated); Study Completion 2028-05-20 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 2 years

SECONDARY OUTCOMES:
Progression - Free Survival（PFS） | Up to 2 years
Minimal Residual Disease - negative rate | Up to 2 years
Number of Participants With Adverse Events and Serious Adverse Events | Up to 2 years
Overall Survival（OS） | Up to 2 years
Duration of Response（DOR） | up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China